CLINICAL TRIAL: NCT03753880
Title: Efficacy of NHS-PEG (Pentaerythirol Polyethylene Glycol Ether Tetra-succinimidyl Glutarate) Coated Collagen Patch (Hemopatch®) for Prevention of Bile Leaks After Liver Resection
Brief Title: Hemopatch for Prevention of Bile Leaks After Liver Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christoph Schwarz, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MUV 1.0
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Bile Leak
Keywords: Liver resection; Bile leaks; Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hemopatch (Experimental): Hemopatch used to cover the resection surface after LR
  Interventions: Device: HEMOPATCH Sealing Hemostat

INTERVENTIONS:
Device: HEMOPATCH Sealing Hemostat — Hemopatch sealing hemostat used after LR to cover the resection surface

SUMMARY:
In liver surgery bile leaks are still a major cause of postoperative morbidity with the need for additional diagnostic tests, additional interventions, prolonged hospital stay, mortality and higher costs. Efforts to further reduce the rate of postoperative biliary morbidity are therefore important.A new polyethylene glycol (PEG)-coated collagen pad (Hemopatch®) showed faster and more sustained hemostasis, less blood loss, and lower hematoma formation than the fibrin-coated collagen patch in an animal model. This might be attributed to an improved tissue adherence of the PEG-coated pad. We hypothesize that this strong adherence to the hepatic resection surface may also serve as a mechanical sealant of bile ducts thus preventing biliary leakage.

To date, there exists no study including a sufficient number of patients to clarify whether sealing of the hepatic resection surface with Hemopatch® can reduce the rate of biliary leaks and data regarding the expected difference in the incidence of biliary complications are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Elective hepatic resection

Exclusion Criteria:

* Minor atypical hepatectomy without a plain cut surface
* Contraindications to the application of Hemopatch®

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Bile leaks | 30 days
  biliary leak is defined as bilirubin concentration in the abdominal drain fluid at least 3 times the serum bilirubin concentration on or after postoperative day 3 or as the need for radiologic or operative intervention resulting from biliary collections or biliary peritonitis

SECONDARY OUTCOMES:
Bleeding | 30 days
  Postoperative bleeding that requires surgical intervention
Abscess | 30 days
  Abscess that requires surgical intervention or percutaneous drainage
Mortalitiy | 30 days
  Overall mortality within 30 days post liver resection

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided